CLINICAL TRIAL: NCT01578512
Title: SPARK a Healthy and Fit Lifestyle
Acronym: SPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK083440
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Face-to-Face (Experimental): 8 sessions of weekly group behavioral weight loss treatment
  Interventions: Behavioral: Face-to-Face
- Web-based (Experimental): Participants receive one group face-to-face session followed by 7 web-based lessons, reporting of key behaviors, and feedback on progress.
  Interventions: Behavioral: Web-based
- Single Session (Active Comparator): Single session behavioral weight loss
  Interventions: Behavioral: Single session

INTERVENTIONS:
Behavioral: Face-to-Face — Face-to-Face behavioral weight loss
  Arms: Face-to-Face
Behavioral: Web-based — Web-based behavioral weight loss
  Arms: Web-based
Behavioral: Single session — The core of behavioral weight loss, including calorie and activity prescriptions, are delivered in a single group treatment session.
  Arms: Single Session

SUMMARY:
The purpose of this study is to determine the best format for delivering a brief behavioral weight loss intervention to young adults 18-25 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 18-25 years old
* body mass index 25-45
* willing to be randomly assigned to any of the 3 arms
* available during the time frame of the study
* willing to complete assessment visits at 0, 2, 4 and 6 months

Exclusion Criteria:

* Age or BMI outside of eligible range
* Medical condition that would interfere with weight loss or make unsupervised physical activity unsafe
* Pregnant or nursing within 6 months
* recent weight loss >10% of body weight
* History of eating disorder
* Substance abuse or dependence

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-08 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Weight | 2 months (post-treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, the Miriam Hospital, Providence, Rhode Island, United States